CLINICAL TRIAL: NCT02681939
Title: Effect of Supplementation of Tulsi (Ocimum Sanctum Linn.) on Metabolic Parameters and Liver Enzymes in Young Overweight and Obese Subjects
Brief Title: Effect of Tulsi (Ocimum Sanctum) on Biochemical Parameters in Young Overweight and Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Sushil Chandra Mahapatra, Professor and Head, Department of Physiology, All India Institute of Medical Sciences, Bhubaneswar, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T/IM-NF/Physio/15/04
Record Dates: First submitted 2016-02-09; First posted 2016-02-15 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tulsi (Experimental): One capsule of Tulsi (Ocimum sanctum) orally, every morning and evening in empty stomach for 60 days regularly.
  Interventions: Drug: Tulsi(Ocimum sanctum Linn.) capsules
- No Tulsi (No Intervention): No intervention

INTERVENTIONS:
Drug: Tulsi(Ocimum sanctum Linn.) capsules
  Arms: Tulsi

SUMMARY:
This is a study to investigate the effect of Tulsi (Ocimum sanctum Linn.) on metabolic and biochemical parameters in young overweight and obese subjects. Thirty overweight/obese volunteers will be divided into two groups. The first group will receive no intervention. The second group will be supplemented with one capsule of Tulsi orally every morning and evening in empty stomach for 60 days. The metabolic parameters and liver enzymes will be evaluated before and after the intervention.

DETAILED DESCRIPTION:
This is a randomized, parallel group, open label pilot study to investigate the effect of Tulsi (Ocimum sanctum Linn.) on metabolic and biochemical parameters in young overweight and obese subjects. Thirty overweight/obese volunteers will be divided into two groups. The first group will receive no intervention. The second group will be supplemented with one capsule of Tulsi orally every morning and evening in empty stomach for 60 days. The metabolic parameters and liver enzymes will be evaluated before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese volunteers of both genders from age 17 to 30 years

Exclusion Criteria:

* Addiction to tobacco and/or alcohol.
* Not on drugs like fluoroquinolones, anticonvulsants, antihypertensives, corticosteroids, hormonal contraceptives, hypolipidemic agents, anti psychotics, protease inhibitors and isotretinoin.
* Not suffering from liver disease, malabsorption, nephrotic syndrome, thyroid disorder, allergy or any other chronic disease.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Serum lipid profile | 60 days

SECONDARY OUTCOMES:
Fasting plasma glucose | 60 days
Fasting plasma insulin | 60 days
Serum liver enzymes | 60 days
Insulin resistance | 60 days
  Using homeostatic model assessment(HOMA2)
Body mass index | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Sushil Ch Mahapatra, MBBS, MD, Principal Investigator — All India Institute of Medical Sciences, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Bhubaneswar, Odisha, India